CLINICAL TRIAL: NCT01409135
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Escalating Doses of AGS-22M6E or ASG-22CE Given as Monotherapy Followed by Expansion Cohorts in Subjects With Malignant Solid Tumors That Express Nectin-4
Brief Title: A Study of the Safety and Pharmacokinetics of AGS-22M6E in Subjects With Malignant Solid Tumors That Express Nectin-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-22M6E-11-1
Record Dates: First submitted 2011-07-29; First posted 2011-08-04 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Tumors; Medical Oncology; Neoplasms
Keywords: Nectin 4 protein, humans; Cancer; Pharmacokinetics of AGS-22M6E; Pharmacokinetics of ASG-22CE; Safety; Clinical Trial, Phase 1; ASG-22ME; AGS-22M6E; ASG-22CE; ASG-22C3
MeSH Terms: conditions — Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- AGS-22M6E-11-1 Dose Level 1 (Experimental)
  Interventions: Drug: AGS-22M6E
- AGS-22M6E-11-1 Dose Level 2 (Experimental)
  Interventions: Drug: AGS-22M6E
- AGS-22M6E-11-1 Dose Level 3 (Experimental)
  Interventions: Drug: AGS-22M6E
- AGS-22M6E-11-1 Dose Level 4 (Experimental)
  Interventions: Drug: AGS-22M6E
- AGS-22M6E-11-1 Dose Level 5 (Experimental)
  Interventions: Drug: AGS-22M6E
- AGS-22M6E-11-1 Dose Level 6 (Experimental)
  Interventions: Drug: AGS-22M6E
- ASG-22CE Expansion Cohort 1 (Experimental): Breast Cancer
  Interventions: Drug: ASG-22CE
- ASG-22CE Expansion Cohort 2 (Experimental): Bladder Cancer
  Interventions: Drug: ASG-22CE
- ASG-22CE Expansion Cohort 3 (Experimental): Lung plus other solid tumor cancers
  Interventions: Drug: ASG-22CE

INTERVENTIONS:
Drug: AGS-22M6E — IV Infusion
  Arms: AGS-22M6E-11-1 Dose Level 1; AGS-22M6E-11-1 Dose Level 2; AGS-22M6E-11-1 Dose Level 3; AGS-22M6E-11-1 Dose Level 4; AGS-22M6E-11-1 Dose Level 5; AGS-22M6E-11-1 Dose Level 6
Drug: ASG-22CE — IV Infusion
  Arms: ASG-22CE Expansion Cohort 1; ASG-22CE Expansion Cohort 2; ASG-22CE Expansion Cohort 3

SUMMARY:
A study examining the safety of AGS-22M6E or ASG-22CE administered as monotherapy therapy in subjects with malignant solid tumors that express Nectin-4.

DETAILED DESCRIPTION:
AGS-22M6E and ASG-22CE are fully human monoclonal antibody conjugated to a cytotoxic agent monomethyl auristatin E (MMAE) targeting Nectin-4 (Agensys code name AGS-22). The main difference between AGS-22M6E and ASG-22CE is the change in cell line for antibody production. AGS-22M6E and ASG-22CE will be administered at mg/kg doses based on the subjects weight at baseline and doses will not change unless the subjects weight changes by ≥ 10% from their baseline weight or the investigational product Dosage Assessment criteria is met.

Subjects will be prescreened for Nectin-4 expression prior to undergoing screening procedures for the main study. Subjects with tumors positive for Nectin-4 expression may be screened for eligibility into the main study. The dose escalation period is estimated to take between 12 and 18 months depending on whether 3 or 6 subjects are enrolled in a given dose cohort, and the availability of consenting subjects.

Subjects will be treated in the dose escalation phase of the study until the maximum tolerated dose (MTD) and recommended dose for expansion (RDE) has been determined by the data review team (DRT). After the RDE has been determined, subjects will be enrolled into 1 of 3 expansion cohorts. There will be 3 expansion cohorts, each targeting a specific cancer (i.e.,Breast, Bladder and Lung plus other solid tumor cancers). The DRT may recommend stopping the study, adjusting the dose or amending the trial at any time.

The clinical bridging to the ASG-22CE involves treating the subjects with ASG-22CE, irrespective of cancer type, at the next lowest dose level previously determined to be safe for AGS-22M6E. After the initial subjects are treated at the bridging dose with ASG-22CE and have completed the safety assessment, future subjects will only be treated with ASG-22CE throughout the remainder of the study.

A disease assessment will be performed by the investigator at Week 8 (± 14 days). Subjects without evidence of disease progression may continue to receive treatment until disease progression or intolerability.

ELIGIBILITY:
Inclusion Criteria: (For Dose Escalation and Dose Expansion)

* Subjects must have a tumor positive for Nectin-4 expression (as measured by central laboratory using primary or metastatic tumor tissue
* Histologically confirmed malignant solid tumors (excluding sarcoma) that have failed all FDA approved therapies indicated for the type of metastatic cancer and line of therapy or for which they were not a candidate to receive treatment
* Measurable disease according to RECIST criteria (version 1.1) (Eisenhauer, et. al.) defined as tumor lesions that are accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

  * 10mm by CT scan (CT scan slice thickness no greater than 5mm
  * 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as nonmeasurable
  * 20 mm by chest X-ray
  * ≥ 15 mm in short axis for lymph nodes when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm)

Note: bone lesions, ascites, and pleural effusions are not considered measurable lesions

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Negative pregnancy test (women of childbearing potential)
* Hematologic function, as follows:

  * a. Absolute neutrophil count (ANC) ≥ 1.0 x109 /L
  * b. Platelet count ≥ 100 x 109/L
  * c. Hemoglobin ≥ 8.5 g/dL
* Renal function, as follows: serum creatinine ≤ 2.0 mg/dL, or measured 24 hour creatinine clearance of ≥ 45 mL/min
* Total bilirubin ≤1.5 x upper limit of normal (ULN)
* Serum albumin > 2.5 g/dL
* Aspartate aminotransferase (AST) ≤ 1.5 x ULN
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN
* Gamma GT ≤1.5 ULN
* International normalized ratio (INR) < 1.5 (or ≤ 3 if on warfarin or other medications for therapeutic anticoagulation)
* Women and men of childbearing potential must be advised and agree to practice effective methods of contraception during the course of the study

Inclusion Criteria for Dose Expansion Only:

In addition to the inclusion criteria listed above, the following criteria will also be required for each expansion cohort:

Expansion Cohort 1: Breast Cancer

* Subjects with Histologically or cytologically diagnosed metastatic breast cancer

Expansion Cohort 2: Bladder Cancer

* Histologically or cytologically confirmed bladder cancer with visceral metastases

Expansion Cohort 3: Lung plus other solid tumor cancer

* Histologically or cytologically confirmed metastatic non-small cell lung cancer (NSCLC) or any other solid tumor cancer

Exclusion Criteria:

* Preexisting neuropathy Grade ≥ 3 or motor neuropathy Grade ≥ 2
* Uncontrolled brain or epidural spinal metastases
* Use of any investigational drug within 14 days or 5 half-lives prior to first dose of study drug
* Any anticancer therapy including: small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy, radiotherapy or any other agents to treat cancer within 28 days prior to first dose of study drug
* Active angina or Class III or IV Congestive Heart Failure (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of the first dose of study drug, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by medication
* Known HIV or AIDS
* Decompensated liver disease as evidenced by clinically significant ascites refractory to diuretic therapy, hepatic encephalopathy, or coagulopathy
* History of thromboembolic events and bleeding disorders ≤ 3 months (e.g.,deep vein thrombosis ( DVT) or pulmonary embolism ( PE)) prior to first dose of study drug
* Major surgery within 28 days prior to first dose of study drug
* Active infection requiring treatment ≤7 days prior to first dose of study drug
* Anti-androgen therapy initiated within 28 days of enrollment (for prostate cancer patients only)
* Positive Hepatitis B surface antigen test
* Positive Hepatitis C antibody test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days after the last dose of study drug
Composite of Pharmacokinetics: Ceoi or Cmax, Ctrough, Tmax, AUC0-21, t½, CL, Vss | Up to 28 days after the last dose of study drug
  Concentration at the end of infusion (Ceoi) or Cmax, trough concentration (Ctrough), Tmax, partial AUC after first dose (AUC0-21), terminal or apparent terminal half-life (t1/2), systemic clearance (CL), volume of distribution at steady state (Vss)

SECONDARY OUTCOMES:
Incidence of anti-drug antibody formation | Up to 28 days after the last dose of study drug
Objective tumor response rate | Every 8 weeks (± 14 days)
  Incidence of a tumor response is defined as a complete or partial response per Response Criteria for Solid Tumors (RECIST version 1.1)
Disease Control Rate | Every 8 weeks (± 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Agensys, Inc.
Locations (9):
- United States (8):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado, Denver-Aurora, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/AGS-22M6E-11-1/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14368&tenant=MT_AST_9011